CLINICAL TRIAL: NCT06085066
Title: The Role of Modified Ultrafiltration on Vascular Resistance, Cardiac Index Enhancement, and Inflammation Reduction Following Open Heart Surgery; A Randomized Clinical Trial
Brief Title: The Role of Modified Ultrafiltration Following Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ratna Farida Soenarto, Consultant, Anestesiologist, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes1000
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Cardiopulmonary bypass; Conventional ultrafiltration; Modified ultrafiltration; Systemic vascular resistance; Pulmonary vascular resistance; Cardiac output index; Interleukin-6

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Ultrafiltration alone on Cardiopulmonary bypass (Active Comparator): Conventional ultrafiltration was used on a cardiopulmonary bypass procedure for patients who underwent open heart surgery
  Interventions: Procedure: Conventional Ultrafiltration alone on Cardiopulmonary bypass
- Conventional Ultrafiltration followed by Modified Ultrafitration on Cardiopulmonary bypass (Active Comparator): Modified ultrafiltration was used following the conventional ultrafiltration on cardiopulmonary bypass procedure for patients who underwent open heart surgery
  Interventions: Procedure: Conventional Ultrafiltration followed by Modified Ultrafitration on Cardiopulmonary bypass

INTERVENTIONS:
Procedure: Conventional Ultrafiltration alone on Cardiopulmonary bypass — Conventional Ultrafiltration was used on Cardiopulmonary bypass for patients who underwent open heart surgery
  Arms: Conventional Ultrafiltration alone on Cardiopulmonary bypass
Procedure: Conventional Ultrafiltration followed by Modified Ultrafitration on Cardiopulmonary bypass — Modified Ultrafiltration was used following the Conventional Ultrafiltration on Cardiopulmonary bypass for patients who underwent open heart surgery
  Arms: Conventional Ultrafiltration followed by Modified Ultrafitration on Cardiopulmonary bypass

SUMMARY:
This study aims to investigate the effect of combining conventional ultrafiltration and modified ultrafiltration compared to conventional ultrafiltration alone in patients who underwent open heart surgery.

DETAILED DESCRIPTION:
The target of this study is adult patients diagnosed with coronary heart disease and valve disease who underwent open heart surgery in CICU PJT RSCM and Jakarta Heart Hospital. The research was conducted after obtaining approval from the FKUI-RSCM ethical committee, and the research subjects agreed to participate by signing an informed consent form. The anesthesia team prepared research subjects undergoing surgery with the placement of arterial cannulas, central venous catheters, sheath introducers, pulmonary artery catheters, and anesthesia management. The placement of these instruments aimed at measuring dependent variables studied included Systemic Vascular Resistance (SVR), Pulmonary Vascular Resistance (PVR), Cardiac Index (CI), and IL-6 levels. The CPB machine was used during the heart chamber opening procedure or coronary artery graft placement, and CUF was initiated. After CPB use was concluded, research subjects were allocated to either the control group or the treatment group through randomization. MUF was performed post-CPB in the treatment group, with the pump speed not exceeding 10% of full flow for 10 minutes. IL-6 levels were measured twice, namely before induction of anesthesia and 24 hours after CPB. SVR, PVR, and CI measurements were carried out before CPB, post-CPB, 10 minutes post-CPB, and 24 hours post-CPB.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older undergoing elective open heart surgery
* Willing to become a research participant and sign an informed consent statement

Exclusion Criteria:

* Patients undergoing redo surgery and emergency surgery
* Patients that have immune disease, chronic lung disease, undergoing hemodialysis
* Patients who are pregnant

Drop-out Criteria

* Patients who experience repeated back-on bypass
* Patients who experience reopen surgery 24 hours after surgery
* Patients who die within 24 hours after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 | 24 hours
  Comparison of IL-6 levels between combination conventional ultrafiltration and modified ultrafiltration with conventional ultrafiltration only on cardiopulmonary bypass. IL-6 levels were assessed using blood samples drawn through a Central Venous Catheter installed before the procedure. Elevated IL-6 levels are indicative of heightened inflammation in the patient, correlating with a more adverse outcome.
Systemic Vascular Resistance (SVR) | 24 hours
  Comparison of SVR between combination conventional ultrafiltration and modified ultrafiltration with conventional ultrafiltration only on cardiopulmonary bypass.
  SVR is the aortic resistance value that the left heart must surpass to pump blood out effectively. SVR measurements are acquired by placing a Pulmonary Artery Catheter in the jugular vein, which is subsequently connected to a Philips monitor. This allows for automatic reading of SVR in dyne.sec/cm5 units through the monitor.
Pulmonary Vascular Resistance (PVR) | 24 hours
  Comparison of PVR between combination conventional ultrafiltration and modified ultrafiltration with conventional ultrafiltration only on cardiopulmonary bypass. PVR is the pulmonary artery resistance value that the right heart must surmount to efficiently pump blood out. PVR measurements are derived from the insertion of a Pulmonary Artery Catheter via the jugular vein, which is subsequently linked to a Philips monitor, facilitating automated readings in units of dyne.sec/cm5 through the monitor.
Cardiac Index | 24 hours
  Comparison of Cardiac Index between combination conventional ultrafiltration and modified ultrafiltration with conventional ultrafiltration only on cardiopulmonary bypass. The cardiac index (CI) represents the volume of blood continuously ejected from the left heart in one minute, relative to the body surface area. CI measurements are acquired through the insertion of a Pulmonary Artery Catheter via the jugular vein, which is subsequently linked to a Philips monitor. This allows for automatic readings in units of L/minute/m2. A higher CI value corresponds to a more favorable patient outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ratna F Soenarto, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmoud AB, Burhani MS, Hannef AA, Jamjoom AA, Al-Githmi IS, Baslaim GM. Effect of modified ultrafiltration on pulmonary function after cardiopulmonary bypass. Chest. 2005 Nov;128(5):3447-53. doi: 10.1378/chest.128.5.3447. PMID 16304298
- [Background] Luciani GB, Menon T, Vecchi B, Auriemma S, Mazzucco A. Modified ultrafiltration reduces morbidity after adult cardiac operations: a prospective, randomized clinical trial. Circulation. 2001 Sep 18;104(12 Suppl 1):I253-9. doi: 10.1161/hc37t1.094931. PMID 11568065
- [Background] Lomivorotov VV, Efremov SM, Kirov MY, Fominskiy EV, Karaskov AM. Low-Cardiac-Output Syndrome After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):291-308. doi: 10.1053/j.jvca.2016.05.029. Epub 2016 Jul 29. No abstract available. PMID 27671216
- [Background] Chandler HK, Kirsch R. Management of the Low Cardiac Output Syndrome Following Surgery for Congenital Heart Disease. Curr Cardiol Rev. 2016;12(2):107-11. doi: 10.2174/1573403x12666151119164647. PMID 26585039
- [Background] Suleiman MS, Zacharowski K, Angelini GD. Inflammatory response and cardioprotection during open-heart surgery: the importance of anaesthetics. Br J Pharmacol. 2008 Jan;153(1):21-33. doi: 10.1038/sj.bjp.0707526. Epub 2007 Oct 22. PMID 17952108
- [Background] Young RW. Prevention of lung injury in cardiac surgery: a review. J Extra Corpor Technol. 2014 Jun;46(2):130-41. PMID 25208430
- [Background] Paparella D, Yau TM, Young E. Cardiopulmonary bypass induced inflammation: pathophysiology and treatment. An update. Eur J Cardiothorac Surg. 2002 Feb;21(2):232-44. doi: 10.1016/s1010-7940(01)01099-5. PMID 11825729
- [Background] Bronicki RA, Hall M. Cardiopulmonary Bypass-Induced Inflammatory Response: Pathophysiology and Treatment. Pediatr Crit Care Med. 2016 Aug;17(8 Suppl 1):S272-8. doi: 10.1097/PCC.0000000000000759. PMID 27490610
- [Background] Zakkar M, Ascione R, James AF, Angelini GD, Suleiman MS. Inflammation, oxidative stress and postoperative atrial fibrillation in cardiac surgery. Pharmacol Ther. 2015 Oct;154:13-20. doi: 10.1016/j.pharmthera.2015.06.009. Epub 2015 Jun 24. PMID 26116810
- [Background] Atkins BZ, Danielson DS, Fitzpatrick CM, Dixon P, Petersen RP, Carpenter AJ. Modified ultrafiltration attenuates pulmonary-derived inflammatory mediators in response to cardiopulmonary bypass. Interact Cardiovasc Thorac Surg. 2010 Nov;11(5):599-603. doi: 10.1510/icvts.2010.234344. Epub 2010 Aug 3. PMID 20682630
- [Background] Sheikhi MA, Ebadi A, Shahriary A, Davoodzadeh H, Rahmani H. Cardiac Surgery Anesthesia And Systemic Inflammatory Response. Int J Bioassays. 2015;4(2):3648-3655. doi: 10.21746/ijbio.2015.02.005. PMID 27857938
- [Background] Muller-Werdan U, Prondzinsky R, Werdan K. Effect of inflammatory mediators on cardiovascular function. Curr Opin Crit Care. 2016 Oct;22(5):453-63. doi: 10.1097/MCC.0000000000000345. PMID 27583586
- [Background] Chew MS, Brix-Christensen V, Ravn HB, Brandslund I, Ditlevsen E, Pedersen J, Hjortholm K, Hansen OK, Tonnesen E, Hjortdal VE. Effect of modified ultrafiltration on the inflammatory response in paediatric open-heart surgery: a prospective, randomized study. Perfusion. 2002 Sep;17(5):327-33. doi: 10.1191/0267659102pf595oa. PMID 12243435
- [Background] Ziyaeifard M, Alizadehasl A, Aghdaii N, Rahimzadeh P, Masoumi G, Golzari SE, Fatahi M, Gorjipur F. The effect of combined conventional and modified ultrafiltration on mechanical ventilation and hemodynamic changes in congenital heart surgery. J Res Med Sci. 2016 Nov 7;21:113. doi: 10.4103/1735-1995.193504. eCollection 2016. PMID 28255321
- [Background] Perez-Vela JL, Ruiz-Alonso E, Guillen-Ramirez F, Garcia-Maellas MT, Renes-Carreno E, Cerro-Garcia M, Cortina-Romero J, Hernandez-Rodriguez I. ICU outcomes in adult cardiac surgery patients in relation to ultrafiltration type. Perfusion. 2008 Mar;23(2):79-87. doi: 10.1177/0267659108095167. PMID 18840575
- [Background] Papadopoulos N, Bakhtiary F, Grun V, Weber CF, Strasser C, Moritz A. The effect of normovolemic modified ultrafiltration on inflammatory mediators, endotoxins, terminal complement complexes and clinical outcome in high-risk cardiac surgery patients. Perfusion. 2013 Jul;28(4):306-14. doi: 10.1177/0267659113478450. Epub 2013 Feb 19. PMID 23429100
- [Background] Onoe M, Magara T, Yamamoto Y, Nojima T. Modified ultrafiltration removes serum interleukin-8 in adult cardiac surgery. Perfusion. 2001 Jan;16(1):37-42. doi: 10.1177/026765910101600106. PMID 11192306